CLINICAL TRIAL: NCT04700488
Title: MRI Imaging to Predict Outcomes of Treatment in PDAC Patients
Brief Title: Magnetic Resonance Imaging (MRI) to Predict Outcomes of Pancreatic Ductal Adenocarcinoma (PDAC)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Cedars-Sinai Cancer Center Protocol Review and Monitoring Committee has requested several protocol modifications and clarifications regarding study outcomes and completion of data entry for subjects who exited the study. Changes are in the process.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Srinivas Gaddam, Associate Director Pancreatic Biliary Research, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000573
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 6D-MRI (Experimental): Participants will undergo 6D-MRI imaging three times throughout the course of the study: once pre-NAT treatment, once during NAT treatment, and once post-NAT treatment.
  Interventions: Diagnostic Test: 6D-MRI

INTERVENTIONS:
Diagnostic Test: 6D-MRI — Six-Dimensional Quantitative Dynamic Contrast Enhanced MRI

SUMMARY:
The purpose of this study is to assess if Six-Dimensional Magnetic Resonance Imaging (6D-MRI) is effective in predicting outcomes in patients with pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
The overarching goal of this pilot study is to evaluate the usefulness of a novel Magnetic Resonance Imaging (MRI) approach, which measure properties of tumor microenvironment (i.e. vascularity, fibrosis), to predict PDAC response to neoadjuvant therapy (NAT).

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer patients (with resectable or borderline resectable or locally advanced tumors) who will undergo neoadjuvant chemotherapy
* Patients able to undergo at least two sets of MRI sessions

Exclusion Criteria:

* Patients who have previously been treated for PDAC
* Patients unable to undergo MRI exam w/contrast
* Patients with metastatic pancreatic cancer visualized on index diagnostic imaging
* Patients with certain metallic implants
* Patients experiencing claustrophobia
* Persons with allergy to animal dander or animal-instigated asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of progression-free survival from baseline | 2 years
  Progression-free survival will be determined by tumor activity assessed from radiomic features on imaging.
Number of participants with R0 resection | 2 years
  The rate of negative tumor resection margins for patient's with resectable cancer that undergo surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pandol, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States